CLINICAL TRIAL: NCT05191589
Title: Haptic Devices vs Non Haptic Devices - Results of a Randomized Trial
Brief Title: Haptic Devices Impact on Laparoscopic Simulators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Anishan Vamadevan, Medical Student and Research Fellow, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAMES
Record Dates: First submitted 2021-02-11; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Medical Education
MeSH Terms: interventions — Haptic Technology

STUDY DESIGN:
Intervention Model Description: Trainees/participants are randomized to either control or interventional group. After reaching proficiency participants must come back after 3-6 weeks to perform a retention test.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the intervention group trainees will train in an already validated laparoscopic training program with haptic devices.
  Interventions: Other: Haptic
- Control (No Intervention): In the control group trainees will complete the same validated training program in the conventional non-haptic setting.

INTERVENTIONS:
Other: Haptic — Trainees are randomized in this group to use the haptic device.
  Arms: Intervention Group

SUMMARY:
The study investigates the impact haptic devices have on reaching proficiency on a laparoscopic simulator as well as investigation if there is a difference in retention of the acquired skills.

ELIGIBILITY:
Inclusion Criteria:

* Must be a junior doctor working in a surgical department

Exclusion Criteria:

* Having performed any laparoscopic surgeries as primary surgeon
* Lack of Basic Danish on a conversational basis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Time (minutes) to reach the predefined proficiency level for the basic skills and salpingectomy procedure | From randomization till participants have passed all modules on the simulator (approx 3-4 weeks)
  Measured in minutes

SECONDARY OUTCOMES:
Time (minutes) to reach the predefined proficiency level for the basic skills and salpingectomy procedure after 3-6 weeks without laparoscopic training on the non-haptic devices (retention test). | From randomization till participants passes all modules on the virtual reality simulator in the trial (approx. 3-4 weeks)
  Measured in minutes

OTHER OUTCOMES:
Exploratory outcome: To observe and register mechanical/technical malfunctions during the intervention and retention. | During trial, up to 1 year
  All mechanical malfunction will be registered and classified afterwards

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - CAMES, Copenhagen, Capital Region
  - CAMES, Copenhagen

IPD SHARING:
Plan to Share IPD: No